CLINICAL TRIAL: NCT07115472
Title: Fluoxetine as a Non-Surgical Intervention for Refractory Superior Mesenteric Artery Syndrome With Comorbid Somatic Symptom Disorder: A Prospective Case Series Study
Brief Title: Fluoxetine in Refractory Superior Mesenteric Artery Syndrome by Targeting Comorbid Somatic Symptom Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhifeng Zhao, PhD, Dr., Xijing Hospital of Digestive Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20242188
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Superior Mesenteric Artery Syndrome; Somatic Symptom Disorder (DSM-5)
Keywords: Fluoxetine
MeSH Terms: conditions — Superior Mesenteric Artery Syndrome | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluoxetine (Experimental): Refractory SMAS patients with SSD received oral fluoxetine treatment, initiated at 20 mg/day and increased to a maximum of 60 mg/day based on therapeutic response.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Refractory SMAS patients with SSD received oral fluoxetine treatment, initiated at 20 mg/day and increased to a maximum of 60 mg/day based on therapeutic response.

SUMMARY:
The goal of this interventional study is to evaluate whether fluoxetine, a selective serotonin reuptake inhibitor (SSRI), can alleviate core symptoms and reduce the need for surgical intervention in patients with refractory superior mesenteric artery syndrome (SMAS) who meet diagnostic criteria for somatic symptom disorder (SSD). The main questions it aims to answer are:

Can fluoxetine improve abdominal symptoms and nutritional status in patients with SMAS and comorbid SSD?

Can psychiatric intervention targeting SSD reduce the likelihood of requiring duodenojejunostomy in refractory SMAS?

Participants will:

Receive oral fluoxetine therapy for a planned treatment duration of 6 months.

Undergo baseline and follow-up assessments including symptom scoring (pain, nausea, dietary intake), body weight/BMI monitoring, and psychiatric evaluation.

Complete psychological questionnaires (PHQ-15, GAD-7, PHQ-9) and resting-state fMRI at baseline and study endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. SMAS was confirmed by two key indicators using imaging or angiographic criteria: aortomesenteric angle of less than 22° or aortomesenteric distance of less than 8 mm;
2. refractory SMAS was defined as failure of conservative treatments, including gastrointestinal decompression, enteral nutrition and parenteral nutrition;
3. accompanied by one or more following characteristics: Severe upper gastrointestinal symptoms (nausea, vomiting, bloating, pain), usually occurring more than once a week; body mass index (BMI)<18.5 kg/m2 related to feeding difficulties;
4. meets the aforementioned criteria for SSD;
5. voluntarily provided informed consent prior to enrollment.

Exclusion Criteria:

1. secondary SMAS due to identifiable causes such as tuberculosis or liver cirrhosis;
2. pregnant or lactating women;
3. patients with malignant tumors or autoimmune diseases;
4. individuals with cardiovascular diseases, organ failure, cognitive impairments, aphasia, or other chronic conditions which interfere with examinations and treatment;
5. psychotropic agents' allergic patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving GOOSS ≥ 2 at 6 months | 6 months after treatment initiation
  Treatment efficacy was evaluated using the Gastric Outlet Obstruction Scoring System (GOOSS), a validated 4-point scale assessing the patient's ability to tolerate oral intake: 0 = no oral intake, 1 = liquids only, 2 = semi-solids, and 3 = low-residue or full diet. The primary efficacy endpoint was the proportion of patients achieving a GOOSS score ≥ 2 at 6 months, indicating the ability to tolerate at least a semi-solid diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact zhaozhifeng@outlook.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: For more information or to submit a request, please contact zhaozhifeng@outlook.com.
URL: https://prsinfo.clinicaltrials.gov/definitions.html